CLINICAL TRIAL: NCT02503995
Title: Influence of Regular Antenatal Physical Exercise on Cardiovascular, Haemodynamic and Autonomic Nervous System (CHANS) Function During and After Pregnancy
Brief Title: Exercise in Pregnancy Evaluative Controlled Study
Acronym: EXPECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swansea University (Other)
Responsible Party: Principal Investigator, Dr Michael Lewis, Associate Professor, Swansea University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 12/WA/0081
Record Dates: First submitted 2015-07-10; First posted 2015-07-21 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- No intervention (Active Comparator): Participants not undertaking any additional exercise
  Interventions: Behavioral: Physical Exercise Participation
- Water-based exercise group (Experimental): Participants assigned to a water-based exercise group
  Interventions: Behavioral: Physical Exercise Participation
- Land-based exercise group (Experimental): Participants assigned to a land-based exercise group
  Interventions: Behavioral: Physical Exercise Participation

INTERVENTIONS:
Behavioral: Physical Exercise Participation

SUMMARY:
This study aimed to investigate whether there are measurable differences in CHANS function in pregnant women who receive only standard antenatal care compared with those who additionally undertake a programme of regular physical exercise.

DETAILED DESCRIPTION:
The health benefits of physical exercise in the non-pregnant population are generally appreciated but its influence during pregnancy has not been clearly demonstrated. The focus of this proposal is to obtain for the first time a comprehensive understanding of the influence of regular physical exercise during pregnancy on cardiovascular, haemodynamic and autonomic nervous system (CHANS) parameters during pregnancy and following childbirth. This will involve assessing heart rate variability and cardiac stroke volume. This study will allow the investigators to compare CHANS parameters in pregnant women who are randomly assigned into three groups: a 'standard care' group and two groups who engage in a supervised programme of physical exercise (either land-based or water-based). The investigators will assess CHANS parameters at three stages during pregnancy and on one occasion following childbirth. This will allow the influence of regular (weekly) physical exercise on CHANS physiology to be assessed during advancing gestation. The investigators will thus use this study to provide initial evidence of the health benefits of regular and specific forms of antenatal physical exercise.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants were apparently healthy pregnant women aged 18 years or over, with no existing complications of pregnancy at their 12-week dating scan.

Exclusion Criteria:

* Exclusion criteria were: a history of cardiovascular or chronic respiratory problems, sleep apnoea, or central/peripheral nervous system disorder.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2012-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability - Time Point 1 | 10-12 weeks gestation
  Determined from 3-lead ECG, assessed as absolute value
Heart Rate Variability - Time Point 2 | 24-28 weeks gestation
  Determined from 3-lead ECG, assessed as absolute value
Heart Rate Variability - Time Point 3 | 34-36 weeks gestation
  Determined from 3-lead ECG, assessed as absolute value
Heart Rate Variability - Time Point 4 | 12 weeks post-birth
  Determined from 3-lead ECG, assessed as absolute value
Cardiac Stroke Volume - Time Point 1 | 10-12 weeks gestation
  Determined from thoracic impedance cardiogram, assessed as absolute value
Cardiac Stroke Volume - Time Point 2 | 24-28 weeks gestation
  Determined from thoracic impedance cardiogram, assessed as absolute value
Cardiac Stroke Volume - Time Point 3 | 34-36 weeks gestation
  Determined from thoracic impedance cardiogram, assessed as absolute value
Cardiac Stroke Volume - Time Point 4 | 12 weeks post-birth
  Determined from thoracic impedance cardiogram, assessed as absolute value

CONTACTS AND LOCATIONS:
Overall Officials: Simon J Emery, MB BCh, Study Director — Abertawe Bro Morgannwg University Health Board

REFERENCES:
- [Result] Carpenter RE, D'Silva LA, Emery SJ, Uzun O, Rassi D, Lewis MJ. Changes in heart rate variability and QT variability during the first trimester of pregnancy. Physiol Meas. 2015 Mar;36(3):531-45. doi: 10.1088/0967-3334/36/3/531. Epub 2015 Feb 18. PMID 25690105
- [Result] D'Silva LA, Davies RE, Emery SJ, Lewis MJ. Influence of somatic state on cardiovascular measurements in pregnancy. Physiol Meas. 2014 Jan;35(1):15-29. doi: 10.1088/0967-3334/35/1/15. Epub 2013 Dec 17. PMID 24345774
- [Derived] Carpenter RE, Emery SJ, Uzun O, D'Silva LA, Lewis MJ. Influence of antenatal physical exercise on haemodynamics in pregnant women: a flexible randomisation approach. BMC Pregnancy Childbirth. 2015 Aug 22;15:186. doi: 10.1186/s12884-015-0620-2. PMID 26296647